CLINICAL TRIAL: NCT01965548
Title: Treatment of Splenic Trauma: a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: Miltstudie1
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Splenic Injury
Keywords: spleen; injury; patient transfer; splenectomy; embolization, theurapeutic
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Splenic injury: All patients admitted at the University Hospital North Norway Tromsø with a splenic injury following trauma, are included in the study.
  Interventions: Procedure: Treatment of splenic injury

INTERVENTIONS:
Procedure: Treatment of splenic injury — There are four possible treatments of splenic injury in this study:
  * splenectomy
  * splenic artery embolisation
  * non-operative management
  * any combination of the three treatments mentioned

SUMMARY:
In blunt trauma, the spleen is most frequent injured organ in the abdomen and the most frequent source of bleeding in the abdomen.

Historically, splenectomy was the treatment of choice for splenic bleeding. For exsanguinating patients, open splenectomy is still the proper choice of treatment if the spleen is a significant source of bleeding. However, for hemodynamic stable patients with splenic injury, non-operative management (NOM) is an alternative, assuming they have no other indication for surgery (peritonitis).

Non-operative management includes observation and/or splenic artery embolisation (SAE), but the indications for observation and SAE varies between trauma centers. The greatest advantage of NOM is the preservation of splenic function.

In the investigators hospital splenic artery embolisation was introduced in 2007. The investigators want to describe the treatment of splenic injuries in their hospital, to see if the number of splenectomies has been recduced after 2007, and to see if SAE has also been used in transferred trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted at UNN Tromsø in the period of 01.01.2000 - 31.12.2013 and with the discharge diagnosis S36.0 Splenic injury (ICD-10)

Exclusion Criteria:

* no injury/coding error
* iatrogenic injury
* transfer >7 days after injury
* >10 days between injury and first hospital admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a traumatic splenic injury admitted at University Hospital North Norway Tromsø
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
type of splenic trauma treatment | 0-7 days
  There are three different treatments of splenic trauma treatment, resulting in four different treatments:
  * splenectomy
  * splenic artery embolization
  * non-operative management
  * any combination of the three treatments

SECONDARY OUTCOMES:
Mortality | 30 days
Length of hospital stay | 1 - 90 days
Length of stay in the intensive care unit | 0 - 90 days
Emergency procedures | 0 - 7 days
  Emergency procedures includes:
  * Chest tube insertion
  * Hemostatic surgery in the abdomen
  * Hemostatic surgery in the pelvis with packing
  * Thoracotomy
  * Primary stabilization of fractures (external fixation)
  * Endotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Trond Dehli, PhD, Principal Investigator — University Hospital og North Norway
Locations (1):
- University Hospital North Norway Tromsø, Tromsø, Norway

REFERENCES:
- [Derived] Dehli T, Bagenholm A, Trasti NC, Monsen SA, Bartnes K. The treatment of spleen injuries: a retrospective study. Scand J Trauma Resusc Emerg Med. 2015 Oct 29;23:85. doi: 10.1186/s13049-015-0163-6. PMID 26514334